CLINICAL TRIAL: NCT05878808
Title: Obsessions and Suicide in Youth With Bipolar 1 Disorder
Brief Title: Obsessions and Suicidality in Youth With Bipolar 1 Disorder
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Riad abd Elgabbar ayoub, Assist professor, Cairo University
Other Study IDs: MS-545- 2021
Record Dates: First submitted 2023-05-18; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Obsessions; Suicide; Bipolar I Disorder; Obsessive-Compulsive Disorder
Keywords: BSSI; DYBOCS; Bipolar disorder
MeSH Terms: conditions — Obsessive Behavior; Suicide; Obsessive-Compulsive Disorder; Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases with ocd
  Interventions: Diagnostic Test: Psychometric assessment
- Cases without ocd
  Interventions: Diagnostic Test: Psychometric assessment

INTERVENTIONS:
Diagnostic Test: Psychometric assessment — Eighty subjects diagnosed with bipolar I disorder were enrolled in this study, subjects were divided according to the presence or absence of OCD to Group A: Bipolar disorder patients with OCD (n = 26), Group B: Bipolar disorder patients without OCD (n = 54). The following scales were applied: Dimensional Yale-Brown obsessive compulsive scale (DYBOCS)- Beck scale for Suicidal ideations (BSSI) - Hamilton depression rating scale (HDRS) and Young mania rating scale (YMRS).

SUMMARY:
Obsessive-compulsive disorder (OCD) is a common co-morbidity with bipolar I disorder, a comorbidity that is known to increase suicide risk. This study aimed to assess the presence of OCD in youth diagnosed with bipolar I disorder & to evaluate the association between OCD and suicide in the same cohort.

Eighty subjects diagnosed with bipolar I disorder were enrolled in this study, subjects were divided according to the presence or absence of OCD to Group A: Bipolar disorder patients with OCD (n = 26), Group B: Bipolar disorder patients without OCD (n = 54). The following scales were applied: Dimensional Yale-Brown obsessive compulsive scale (DYBOCS)- Beck scale for Suicidal ideations (BSSI) - Hamilton depression rating scale (HDRS) and Young mania rating scale (YMRS).

The results revealed that DYBOCS score of group A was 30.23±0.43, & of group B was 18.50±1.88 with a significant difference (p<0.01). There was a significantpositive correlation between BSSI and age, age of onset and YMRS in Group A (p<0.01).

The study demonstrated that OCD is a common comorbidity in youth with bipolar I disorder and may be associated with a greater risk of suicide than in youth with bipolar I disorder without co-morbid OCD. Furthermore, co-morbidity of OCD with bipolar I disorder in youth may be associated with younger age of onset and more severe symptoms profile.

ELIGIBILITY:
Inclusion Criteria:

- Can read and write, agreed to sign the consent, diagnosed with bipolar I disorder

Exclusion Criteria:

* refused to sign the consent, active manic phase, recent substance use

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Eighty subjects diagnosed with bipolar I disorder were enrolled in this study, subjects were divided according to the presence or absence of OCD to Group A: Bipolar disorder patients with OCD (n = 26), Group B: Bipolar disorder patients without OCD (n = 54).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
Association of OCD with bipolar I disorder | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No